CLINICAL TRIAL: NCT00898313
Title: Molecular Predictors of Lung Cancer Behavior
Brief Title: Molecular Predictors of Cancer in Patients at High Risk of Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fabien Maldonado, Professor of Medicine and Thoracic Surgery, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC THO 0398; P30CA068485 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Comparative Genomic Hybridization; Oligonucleotide Array Sequence Analysis; Blood Specimen Collection; Urine Specimen Collection; Thoracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, nasal cells, sputum, bronchal epithelial cells, airway tissue, and lung tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sample Collection
  Interventions: Genetic: comparative genomic hybridization; Genetic: gene expression microarray analysis; Genetic: proteomic profiling analysis; Other: biologic sample preservation procedure; Procedure: nasal brushing; Procedure: Blood draw; Procedure: Urine collection; Procedure: sputum sample; Procedure: fluorescence bronchoscopy with airway biopsy; Procedure: fine needle aspiration of the lung; Procedure: thoracentesis

INTERVENTIONS:
Genetic: comparative genomic hybridization — Collection of sputum, blood, urine, and a small amount of lung tissue.
Genetic: gene expression microarray analysis — Collection of sputum, blood, urine, and a small amount of lung tissue.
Genetic: proteomic profiling analysis — Collection of sputum, blood, urine, and a small amount of lung tissue.
Other: biologic sample preservation procedure — Collection of sputum, blood, urine, and a small amount of lung tissue.
Procedure: nasal brushing — Using a brush, superficial cells are removed from the nose.
Procedure: Blood draw — Venous blood will be collected
Procedure: Urine collection — Subjects will be asked to provide a urine specimen.
Procedure: sputum sample — Prior to their bronchoscopy, subjects will be asked for a sputum specimen. This is a collection of mucous that you cough up.
Procedure: fluorescence bronchoscopy with airway biopsy — A flexible tube attached to a fluorescent light source will be inserted into the subject's mouth or nose to reach the airway. Samples of the lining of the airway will be taken, as well as bronchial secretions and epithelial cell from brushings of the lining of the airway.
Procedure: fine needle aspiration of the lung — A small needle is inserted into the lung to collect tissue. This procedure will only be performed if the patient's physician orders it.
Procedure: thoracentesis — A small needle is inserted into the patient's lung cavity and a small amount of fluid is collected. This procedure will only be performed if the patient's physician orders it.

SUMMARY:
RATIONALE: Using samples of blood, urine, sputum, and lung tissue from patients at high risk of cancer for laboratory studies may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at molecular predictors of cancer in patients at high risk of lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To use fixed lung tissue for histological evaluation and fresh tissue samples for molecular studies to study DNA, RNA, and protein abnormalities in lung preneoplastic and neoplastic lesions.
* To use proteomic techniques, including matrix-assisted laser desorption ionization-mass spectrometry (MALDI-MS), to develop a method of diagnosing and staging both pre-invasive and invasive lesions, using less invasive methods.

OUTLINE: Blood, urine, nasal cell, and sputum samples are collected. Lung tissue samples are also collected using fluorescence bronchoscopy and epithelial cell collection.

Samples are studied by genetic and proteomic analyses, including comparative genomic hybridization, expression microarray, and protein profiling.

ELIGIBILITY:
Inclusion Criteria:

-All adults referred to Vanderbilt Medical Center, Veterans Administration Medical Center, St. Thomas Hospital and Meharry Medical Center for evaluation of signs or symptoms of lung cancer.

Exclusion Criteria:

* Inability to provide informed consent
* Minors
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who may have lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2003-12; Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
To quantitate the molecular changes during lung cancer development | After collection of designated samples
  As a part of the study nasal brushing specimens, sputum, blood, urine, and a small amount of other tissue will be collected during standard of care procedures (bronchial epithelial, trans-thoracic fine needle aspiration (FNA) and thoracentesis as part of patient work up.
  Clinical diagnosis is the primary goal of the procedure. All the research specimens are collected after the primary goal of the procedure is met.

SECONDARY OUTCOMES:
Develop a method to diagnose and stage pre-invasive and invasive lesions | After collection of designated samples
  Use of proteomic techniques in the laboratory to find a method of diagnosing lung tissue as benign or malignant rather than relying on invasive open-chest surgery for a diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Maldonado, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/